CLINICAL TRIAL: NCT02574676
Title: Prospective Observational Study Measuring the Short-Form36 ( SF-36v2) and Other QOL Tools in an AL Amyloidosis Population
Brief Title: Quality of Life (QOL) Registry for Patients With AL Amyloidosis
Status: Completed | Type: Observational
Sponsor: Prothena Biosciences Ltd. (Industry)
Collaborators: Amyloidosis Research Consortium (Other); Amyloidosis Support Groups (Other); Amyloidosis Foundation (Other); Quality Metrics (Unknown)
Responsible Party: Sponsor
Other Study IDs: CO-083252
Record Dates: First submitted 2015-10-05; First posted 2015-10-14 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: AL Amyloidosis; Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: non-interventional

SUMMARY:
This is an online registry to document the psychometric properties of SF-36v2 among patients with AL Amyloidosis, to document patients' burden of disease, to better understand the patient's experience and to follow quality of life issues using a variety of QOL measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have AL Amyloidosis

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Al Amyloidosis
Sampling Method: Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2015-10; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Psychometric evaluation of short-form 36 (SF-36v2) in patients with AL Amyloidosis | Change from Baseline to 12 months

SECONDARY OUTCOMES:
Calculate burden of illness from participants using SF-36 Mental Component Score (MCS) and Physical Component Score (PCS) compared with sample from US general population and three other chronic conditions: Congestive Heart Failure, Lymphoma and COPD | Baseline- cross sectional
  The comparison is made to other populations from the baseline cross-sectional measurements. There is no timeframe, except baseline
Assess the pathway to diagnosis and treatment through a disease history specific questionnaire collecting organ involvement, initial symptoms, diagnosis duration, treatment received and other disease characteristics | Baseline- cross sectional
  The analysis is done atbaseline .
Psychometric evaluation of Kansas City Cardiomyopathy Questionnaire (KCCQ-12) in patients with AL Amyloidosis | Change from Baseline to 12 months
Psychometric evaluation of Patient Global Impression-Severity Scale (PGI-S) in patients with AL Amyloidosis | Change from Baseline to 12 months
Psychometric evaluation of Patient Global Assessment of Functioning (GAF) Scale in patients with AL Amyloidosis | Change from Baseline to 12 months
Psychometric evaluation of Hematology Patient Reported Symptom Screen (HPRSS) in patients with AL Amyloidosis | Change from Baseline to 12 months
Psychometric evaluation of Work Productivity and Activity Questionnaire: Specific Health Problem V2.0 (WPAI:SHP) in patients with AL Amyloidosis | Change from Baseline to 12 months
Psychometric evaluation of MOS 6-Item Sleep Scale Standard in patients with AL Amyloidosis | Change from Baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Online registry, South San Francisco, California, United States

REFERENCES:
- [Derived] Bayliss M, McCausland KL, Guthrie SD, White MK. The burden of amyloid light chain amyloidosis on health-related quality of life. Orphanet J Rare Dis. 2017 Jan 19;12(1):15. doi: 10.1186/s13023-016-0564-2. PMID 28103898